CLINICAL TRIAL: NCT06500351
Title: Renalase(rs10887800) Genotyping & Leucocytes Telomere Length in Patients With Postpartum Hypertension.
Brief Title: Renalase(rs10887800) Genotyping & Leucocytes Telomere Length in Postpartum. Hypertension
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amera Morad Foad, Assistant Professor of Medical Biochemistry, Sohag University
Other Study IDs: Soh-Med-24-06-08PD
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Renalase(rs10887800) Genotyping & Leucocytes Telomere Length in Patients With Postpartum Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- denovo postpartum hypertension: females with new onset hypertension after delivary
- persitant postpartum hypertension: females with preexisting hypertension or preeclampsia that persist after delivery
- control: females with normal postpartum blood pressure

SUMMARY:
This is an observertional study aimed at Study the association between Renalase(rs10887800) Genotyping & Leucocytes telomere length in patients with postpartum hypertension whether new onset( denovo) or persistent following pregnancy complicated by hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are18 years or above, and have a diagnosis of postpartum hypertension(regardless of where they received their antenatal care) attended to Sohag university hospitals

Exclusion Criteria:

* All pregnant women with medical disorders in pregnancy other than Hypertensive disorders during pregnancy (e.g., sickle cell disease, heart disease, kidney and other connective tissues disorders) will be excluded from the study. Also we excluded measurements taken during scheduled or unscheduled surgical encounters given potential for interaction with anesthetic agents

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — only females are eligible for this study because of its relation to pregnancy.
Study Population: Patients who were 18 years or above, and have a diagnosis of postpartum hypertension
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-06-25 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Renalase(rs10887800) Genotyping | 1 year
  The presence of gene polymorphism whether homogenetic or heterogenetic

SECONDARY OUTCOMES:
Leucocytes telomere length | 1 year
  Measurement of the relative length of WBCs telomere in patints with postpartum hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Amera Morad Foad, assistant professor, Principal Investigator — Sohag University
Locations (1):
- Sohag university hosoital, Sohag, Egypt